CLINICAL TRIAL: NCT00666562
Title: A Phase II Randomized, Placebo-Controlled Trial of Polyphenon E to Evaluate Bladder Tissue Levels of EGCG
Brief Title: Green Tea Extract in Treating Patients With Nonmetastatic Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00906; NCI-2009-00906 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CO06810; CDR0000594276; H-2007-0250; UWI06-8-01 (Other: University of Wisconsin Hospital and Clinics); UWI06-8-01 (Other: DCP); N01CN35153 (NIH); P30CA014520 (NIH)
Record Dates: First submitted 2008-04-24; First posted 2008-04-25 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Stage I Bladder Cancer; Stage II Bladder Cancer; Stage III Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — polyphenon E

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Arm I (placebo) (Placebo Comparator): Patients receive six oral placebo capsules once daily for 14-28 days.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Placebo
- Arm II (polyphenon E, placebo) (Experimental): Patients receive four oral polyphenon E capsules and two oral placebo capsules once daily for 14-28 days in the absence of unacceptable toxicity.
  Interventions: Dietary Supplement: Defined Green Tea Catechin Extract; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Placebo
- Arm III (polyphenon E, trans-urethral resection or cystectomy) (Experimental): Patients receive six oral polyphenon E capsules once daily for 14-28 days in the absence of unacceptable toxicity. After completion of study treatment, patients undergo trans-urethral resection of bladder tumor or cystectomy.
  Interventions: Dietary Supplement: Defined Green Tea Catechin Extract; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Dietary Supplement: Defined Green Tea Catechin Extract — Given orally
  Other Names: Polyphenon E; Polyphenon E TM
  Arms: Arm II (polyphenon E, placebo); Arm III (polyphenon E, trans-urethral resection or cystectomy)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Placebo — Given orally
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm I (placebo); Arm II (polyphenon E, placebo)
Procedure: Therapeutic Conventional Surgery — Undergo surgery
  Arms: Arm III (polyphenon E, trans-urethral resection or cystectomy)

SUMMARY:
Green tea extract contains ingredients that may slow the growth of certain cancers. It is not yet known whether green tea extract is more effective than a placebo when given before surgery in treating patients with bladder. This randomized phase II trial is studying green tea extract to see how well it works compared to a placebo when given before surgery in treating patients with nonmetastatic bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To compare the levels of epigallocatechin-3-gallate (EGCG) in nonmalignant bladder tissue from patients with bladder cancer treated with oral polyphenon E 800 mg EGCG or polyphenon E 1200 mg EGCG once daily for 14-28 days.

SECONDARY OBJECTIVES:

I. To compare the levels of EGCG in nonmalignant versus malignant bladder tissue samples from these patients.

II. To examine the dose-response modulation of surrogate intermediate endpoint biomarkers (e.g., Proliferating Cell Nuclear Antigen [PCNA], Matrix Metallopeptidase 2 [MMP2], clusterin, Vascular endothelial Growth Factor [VEGF], p27, and ODC) in malignant and nonmalignant samples of bladder tissue from these patients after administration of polyphenon E.

III. To correlate EGCG levels in samples of serum, urine, and tissue from these patients.

IV. To examine the levels of other catechins (i.e., epicatechin, epicatechin gallate, and epigallocatechin) found in polyphenon E in samples of serum, urine, and tissue from these patients.

V. To compare the metabolism of EGCG by Catechol-O-Methyltransferase (COMT) and Uridinediphosphate-Glucuronosyltransferase (UGT) in relation to pharmacogenetic polymorphisms in COMT and UGT in samples of serum, urine, and tissue from these patients.

VI. To examine the changes in serum Insulin Growth Factor 1 (IGF-1) and IGFBP-3 levels after administration of polyphenon E in these patients.

OUTLINE:

This is a multicenter study. Patients are stratified according to tumor site and disease invasiveness (invasive vs noninvasive). Patients are randomized to 1 of 3 treatment arms.

Arm I: Patients receive six oral placebo capsules once daily for 14-28 days in the absence of unacceptable toxicity.

Arm II: Patients receive four oral polyphenon E capsules and two oral placebo capsules once daily for 14-28 days in the absence of unacceptable toxicity.

Arm III: Patients receive six oral polyphenon E capsules once daily for 14-28 days in the absence of unacceptable toxicity.

After completion of study treatment, patients undergo trans-urethral resection of bladder tumor or cystectomy.

Blood, urine, and tissue samples are obtained at baseline and at the end of study treatment for correlative laboratory studies. Samples are evaluated for pharmacokinetics of polyphenon E using high performance liquid chromatography. Levels of epigallocatechin-3-gallate [EGCG] and other catechins found in polyphenon E are assessed for correlation in serum, urine, and tissue. Intermediate endpoint biomarkers are evaluated for dose-response modulation in serum (i.e., IGF-1 and IGFBP-3) via ELISA and in bladder tissue obtained at the time of bladder surgery (i.e., PCNA, MMP2, clusterin, VEGF, p27, and ODS) via IHC. Patients at the University of Wisconsin undergo additional biopsy of bladder tissue for matrix-assisted laser desorption quadrupole time-of-flight (O-MALDI-qTOF) analysis of EGCG pharmacokinetics. Tissue samples are examined for intracellular concentration and distribution of EGCG. Genotyping studies for pyrosequencing of UGT and COMT polymorphisms are also performed.

ELIGIBILITY:
Criteria:

* Diagnosis of bladder cancer
* Bladder tumor discovered on cystoscopy within the past 60 days
* Invasive or non-invasive tumor
* Primary tumor may represent either an initial diagnosis or recurrent disease of any clinical stage
* No metastatic disease
* Must be an eligible candidate for a partial cystectomy, radical cystectomy, or trans-urethral resection of bladder tumor (TURBT)
* Has not undergone any treatment for superficial or invasive bladder cancer since the diagnostic cystoscopy
* TURBT or radical cystectomy is the planned curative surgical treatment
* ECOG performance status (PS) 0-1 OR Karnofsky PS 70-100%
* More than 30 days since any prior intravesical therapy or adjuvant chemotherapy
* More than 30 days since prior bladder surgery
* Biopsies are not considered surgeries
* No prior pelvic radiotherapy
* No concurrent systemic chemotherapy for any other cancer, except nonmelanoma skin cancer
* No concurrent NSAIDs (e.g., ibuprofen, naproxen, or cyclooxygenase-2 inhibitors) except =< 81 mg aspirin per day
* Concurrent acetaminophen (Tylenol) or prescription opioids combined with acetaminophen (i.e., Percocet, Darvocet, Vicodin, Tylenol #3) allowed for pain
* No other concurrent investigational agents
* White Blood Cell (WBC) >= 3,000/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 10 g/dL
* Alkaline phosphatase =< upper limit of normal (ULN)
* Bilirubin =< ULN
* Asparate Aminotransferase (AST) and Alanine Transaminase (ALT) =< ULN
* Sodium 135-144 mmol/L (inclusive)
* Potassium 3.2-4.8 mmol/L (inclusive)
* Chloride 85-114 mmol/L (inclusive)
* Bicarbonate >11 mEQ/dL
* Negative pregnancy test
* Fertile patients must use effective contraception
* Willing to avoid green tea beverages and green tea-containing products during study participation
* No evidence of other cancers, except nonmelanoma skin cancer
* No history of allergic reactions attributed to tea or to any of the compounds of similar chemical or biologic composition to Polyphenon E or any of the inactive ingredients in Polyphenon E capsules
* No uncontrolled intercurrent illness including, but not limited to, any of the following: Ongoing or active infection, Symptomatic congestive heart failure, Unstable angina pectoris, Cardiac arrhythmia, Psychiatric illness/social situations that would limit study compliance
* More than 24 hours since prior and no concurrent consumption of any other green tea supplements or more than 2 cups (16 oz) of green tea either through dietary sources or through nutritional supplementation
* Topical cosmetics (i.e., lotions, shampoos, makeup) that contain green tea are allowed
* Creatinine normal
* Not pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-07-02 (Actual); Primary Completion 2012-04-26 (Actual); Study Completion 2017-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Downs, Principal Investigator — University of Wisconsin, Madison
Locations (6):
- United States (6):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - University of Rochester, Rochester, New York
  - Urology San Antonio Research PA, San Antonio, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited during a 4 year period by staff at 5 participating institutions (both University hospitals and community clinics).
Groups:
- Arm I (Placebo): Patients receive six oral placebo capsules once daily for 14-28 days. After completion of study treatment, patients undergo trans-urethral resection of bladder tumor or cystectomy.
  placebo: Given orally
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Arm II (800mg Polyphenon E, Placebo): Patients receive four oral 800mg polyphenon E capsules and two oral placebo capsules once daily for 14-28 days in the absence of unacceptable toxicity.After completion of study treatment, patients undergo trans-urethral resection of bladder tumor or cystectomy.
  defined green tea catechin extract: Given orally
  placebo: Given orally
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Arm III (1200mg Polyphenon E): Patients receive six oral 1200mg polyphenon E capsules once daily for 14-28 days in the absence of unacceptable toxicity. After completion of study treatment, patients undergo trans-urethral resection of bladder tumor or cystectomy.
  defined green tea catechin extract: Given orally
  therapeutic conventional surgery: Undergo surgery
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Started | 11 | 10 | 10
Completed | 11 | 8 | 10
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Concomitant Medication | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E) | Total
Number analyzed (Participants) | 11 | 10 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 3 | 13
  >=65 years | 8 | 3 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.00 (7.04) | 65.20 (9.50) | 66.20 (9.55) | 67.23 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 9 | 9 | 8 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 7
  Not Hispanic or Latino | 8 | 8 | 8 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 11 | 10 | 9 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Epigallocatechin Gallate (EGCG) Levels in Nonmalignant Bladder Tissue (e.g., Normal-appearing Urothelium, Inflammatory Lesions in the Bladder, Sessile Noninvasive Bladder Tumors, and Papillary Noninvasive Bladder Tumors)
Description: Comparison of nonmalignant bladder tissue levels of EGCG between the placebo group and the EGCG groups combined using student t-test.
Time Frame: up to 28 days
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 9 | 8 | 8
ng/mL | 0.00 (0.00) | 0.50 (1.42) | 1.72 (3.11)
Statistical Analysis 1: Comparison: Arm I (Placebo) vs Arm II (800mg Polyphenon E, Placebo) vs Arm III (1200mg Polyphenon E); Test type: Superiority or Other; p = 0.046, t-test, 2 sided

2. Secondary Outcome: Levels of EGCG in Malignant Bladder Tissue
Time Frame: up to 28 days
Population: Analysis was not able to be completed for 1 participant in Arm I, 1 participant in Arm II, and 3 participants in Arm III.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 10 | 7 | 7
ng/mL | 0.00 (0.00) | 0.00 (0.00) | 2.54 (2.92)

3. Secondary Outcome: Levels of Surrogate Intermediate Endpoint Biomarkers in Malignant and Nonmalignant Bladder Tissue Assessed by Immunohistochemistry
Time Frame: up to 28 days
Measure: Mean (Standard Deviation); unit: optical density
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 11 | 8 | 10
optical density
  PCNA | 0.41 (0.052) | 0.38 (0.061) | 0.35 (0.052)
  MMP2 | 0.16 (0.026) | 0.18 (0.054) | 0.16 (0.069)
  Clusterin | 0.074 (0.032) | 0.061 (0.020) | 0.046 (0.013)
  VEGF | 0.011 (0.0065) | 0.021 (0.0173) | 0.013 (0.0066)
  p27 | 0.36 (0.080) | 0.35 (0.090) | 0.31 (0.057)

4. Secondary Outcome: Serum Insulin Growth Factor-1 (IGF-1) Levels Assessed by ELISA
Time Frame: Baseline and up to day 28
Population: Analysis was not able to be completed for 2 participants in Arm I.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 9 | 8 | 10
ng/mL
  Baseline | 135.06 (22.64) | 122.22 (37.49) | 132.12 (15.12)
  End of Study | 131.86 (15.59) | 124.22 (38.06) | 132.27 (27.77)

5. Secondary Outcome: Levels of Other Catechins (Epicatechin Gallate, Epicatechin, and Epigallocatechin) Found in Polyphenon E Tumor Tissue Samples
Time Frame: up to 28 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 10 | 7 | 7
ng/mL
  epicatechin gallate (ECG) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  epicatechin (EC) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  epigallocatechin (EGC) | 0.00 (0.00) | 0.00 (0.00) | 0.60 (1.58)

6. Secondary Outcome: Absolute Change for Baseline From EGCG in Serum Samples
Description: The difference between the amount at the end of study (up to 28 days) from baseline.
Time Frame: Baseline and up to 28 days
Population: Analysis was not able to be completed for 2 participants in Arm I and 1 participant in Arm II.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 9 | 7 | 10
ng/mL | 0.28 (1.11) | 82.33 (83.66) | 85.37 (76.34)

7. Secondary Outcome: Metabolism of EGCG in Serum and Urine in Relation to Pharmacogenetic Polymorphisms in Catechol-O-Methyltransferase (COMT)
Time Frame: At Baseline
Population: This outcome was assessed in all participants,combined irrespective of their randomization.
  Analysis was not able to be completed on 4 participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Glycine/Glycine: G to G transition in the COMT gene
- Alanine/Glycine: A to G transition in the COMT gene
- Alanine/Alanine: A to A transition in the COMT gene
Arm/Group | Glycine/Glycine | Alanine/Glycine | Alanine/Alanine
Number analyzed (Participants) | 6 | 11 | 8
ng/mL
  Plasma | 4.12 (4.80) | 0.57 (1.89) | 2.48 (3.48)
  Serum | 0.00 (0.00) | 0.69 (1.82) | 0.43 (1.21)

8. Secondary Outcome: Serum IGFBP-3 Levels Assessed by ELISA
Time Frame: Baseline and up to 28 days
Population: Analysis was not able to be completed for 2 participants in Arm I.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 9 | 8 | 10
ng/mL
  Baseline | 1918.31 (607.16) | 1679.61 (556.59) | 1824.86 (559.58)
  End of Study | 2020.31 (701.46) | 1800.08 (490.92) | 1624.03 (611.89)

9. Secondary Outcome: Levels of Other Catechins (Epicatechin Gallate, Epicatechin, and Epigallocatechin) Found in Polyphenon E Normal Tissue Samples
Time Frame: up to 28 days
Population: Analysis was not able to be completed for 2 participants in Arm I and 2 participants in Arm III.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 9 | 8 | 8
ng/mL
  epicatechin gallate (ECG) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  epicatechin (EC) | 0.00 (0.00) | 0.00 (0.00) | 0.20 (0.55)
  epigallocatechin (EGC) | 0.00 (0.00) | 0.20 (0.55) | 0.00 (0.00)

10. Secondary Outcome: Absolute Change From Baseline of Other Catechins (Epicatechin Gallate, Epicatechin, and Epigallocatechin) Found in Polyphenon E in Urine Samples
Description: The difference between the amount at the end of study (up to 28 days) from baseline.
Time Frame: Baseline and up to 28 days
Population: Analysis was not able to be completed for 3 participants in Arm I and 1 participant in Arm II.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 8 | 7 | 10
ng/mL
  epicatechin gallate (ECG) | 0.00 (0.00) | 1.13 (1.78) | 1.49 (2.13)
  epicatechin (EC) | 0.52 (1.46) | 2.41 (3.15) | 5.33 (6.78)
  Epigallocatechin (EGC) | 0.20 (0.55) | 3.60 (3.21) | 12.16 (11.09)

11. Secondary Outcome: Absolute Change From Baseline of Other Catechins (Epicatechin Gallate, Epicatechin, and Epigallocatechin) Found in Polyphenon E Plasma Samples
Description: The difference between the amount at the end of study (up to 28 days) from baseline.
Time Frame: Baseline and up to 28 days
Population: Analysis was not able to be completed for 2 participants in Arm I and 1 participant in Arm II.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 9 | 7 | 10
ng/mL
  epicatechin gallate (ECG) | 0.17 (0.52) | 8.38 (11.03) | 8.62 (9.14)
  epicatechin (EC) | 0.00 (0.00) | 0.97 (1.97) | 0.31 (0.66)
  epigallocatechin (EGC) | 0.00 (0.00) | 6.93 (10.06) | 3.46 (4.04)

12. Secondary Outcome: Absolute Change for Baseline of EGCG in Urine Samples
Description: The difference between the amount at the end of study (up to 28 days) from baseline.
Time Frame: Baseline and up to 28 days
Population: Analysis was not able to be completed for 3 participants in Arm I and 1 participant in Arm II.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Number analyzed (Participants) | 8 | 7 | 10
ng/mL | 0.00 (0.00) | 1.93 (0.98) | 3.38 (1.60)

13. Secondary Outcome: Metabolism of EGCG in Serum and Urine in Relation to Pharmacogenetic Polymorphisms in Uridinediphosphate- Glucuronosyltransferase (UGT)
Time Frame: At Baseline
Population: This outcome was assessed in all participants,combined irrespective of their randomization. Analysis was not able to be completed for 4 participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 5/6 Genotype; 6/6 Genotype; 6/7 Genotype; 7/7 Genotype: Genotype of the UGT in EGCG
Arm/Group | 5/6 Genotype | 6/6 Genotype | 6/7 Genotype | 7/7 Genotype
Number analyzed (Participants) | 2 | 7 | 15 | 1
ng/mL
  Plasma | 2.97 (4.20) | 2.09 (3.75) | 2.02 (3.58) | 0.00 (0.00)
  Urine | 1.72 (2.43) | 0.86 (2.27) | 0.10 (0.40) | 0.00 (0.00)

ADVERSE EVENTS:
Arm/Group | Arm I (Placebo) | Arm II (800mg Polyphenon E, Placebo) | Arm III (1200mg Polyphenon E)
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/11 | 5/10 | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Placebo) (N=11) | Arm II (800mg Polyphenon E, Placebo) (N=10) | Arm III (1200mg Polyphenon E) (N=10)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
heartburn (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausa (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
taste alteration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
imb (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (4) | 1 (1)
anal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
extremity limb pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
headache (General disorders) | 0 (0) | 1 (1) | 4 (4)
joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (3)
kidney pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
pelvis pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less